CLINICAL TRIAL: NCT03261778
Title: Conservative Treatment of Rockwood Type III Acromioclavicular Dislocation With Two Different Types of Braces: a Comparative Prospective Randomized Trial
Brief Title: Comparison of Two Types of Braces in the Treatment of Rockwood Type III AC-dislocations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bürgerspital Solothurn (Other)
Collaborators: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Michael Finsterwald, Dr. med. Michael Finsterwald, Bürgerspital Solothurn
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-00670
Record Dates: First submitted 2017-08-18; First posted 2017-08-25 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Acromioclavicular Joint Dislocation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acromion 2.0 Brace (Experimental)
  Interventions: Device: Acromion 2.0 Brace
- Mitella Sling (Active Comparator)
  Interventions: Device: Acromion 2.0 Brace

INTERVENTIONS:
Device: Acromion 2.0 Brace — Acromion 2.0 Brace will be worn for 6 weeks instead of the conventional Mitella sling

SUMMARY:
In a randomised prospective comparative Trial the investigators aim to compare the conservative Treatment of acromioclavicular dislocations (Rockwood III) with a conventional sling versus a Acromion 2.0 brace, which exerts a direct Reposition force on the Joint.

The sling/brace will be worn for 6 weeks and the patients will be regularly checked clinically and radiologically.The investigators are interested in differences of shoulder function, Patient satisfaction as well as cosmetic and radiological results.

ELIGIBILITY:
Inclusion Criteria:

* First acute acromioclavicular dislocation Rockwood Type III

Exclusion Criteria:

* Previous injury to acromioclavicular Joint
* Previous surgery of acromioclavicular Joint
* Known hypersensitivity or allergy to fabric of investigational product
* Pregnancy
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-12 (Actual)

PRIMARY OUTCOMES:
Shoulder function | at 6 weeks
  Constant-Score
Shoulder function | at 12 weeks
  Constant-Score
Shoulder function | at 1 week
  ASES-Score (American Shoulder and Elbow Score)
Shoulder function | at 6 weeks
  ASES-Score (American Shoulder and Elbow Score)
Shoulder function | at 12 weeks
  ASES-Score (American Shoulder and Elbow Score)
Shoulder function | at 1 week
  Subjective Shoulder value (scale 0-100% where 100% equals a healthy shoulder)
Shoulder function | at 6 weeks
  Subjective Shoulder value (scale 0-100% where 100% equals a healthy shoulder)
Shoulder function | at 12 weeks
  Subjective Shoulder value (scale 0-100% where 100% equals a healthy shoulder)

SECONDARY OUTCOMES:
Degree of lateral clavicle dislocation | at initial presentation
  Coracoclavicular distance on Panorama view in comparison to healthy side
Degree of lateral clavicle dislocation | at 6 weeks
  Coracoclavicular distance on Panorama view in comparison to healthy side
Degree of lateral clavicle dislocation | at 12 weeks
  Coracoclavicular distance on Panorama view in comparison to healthy side

CONTACTS AND LOCATIONS:
Overall Officials: Näder Helmy, PD, MD, Study Chair — Bürgerspital Solothurn, Department of Orthopaedics and Traumatology
Locations (2):
- Switzerland (2):
  - Orthopädische Universitätsklinik Basel, Basel
  - Bürgerspital Solothurn, Department of Orthopaedics and Traumatology, Solothurn

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Phillips AM, Smart C, Groom AF. Acromioclavicular dislocation. Conservative or surgical therapy. Clin Orthop Relat Res. 1998 Aug;(353):10-7. PMID 9728155
- [Background] Korsten K, Gunning AC, Leenen LP. Operative or conservative treatment in patients with Rockwood type III acromioclavicular dislocation: a systematic review and update of current literature. Int Orthop. 2014 Apr;38(4):831-8. doi: 10.1007/s00264-013-2143-7. Epub 2013 Oct 31. PMID 24178060
- [Background] Smith TO, Chester R, Pearse EO, Hing CB. Operative versus non-operative management following Rockwood grade III acromioclavicular separation: a meta-analysis of the current evidence base. J Orthop Traumatol. 2011 Mar;12(1):19-27. doi: 10.1007/s10195-011-0127-1. Epub 2011 Feb 23. PMID 21344264
- [Derived] Duffett RW, Duralde XA, Marcus RE. CORR Synthesis: What Is the Most Effective Treatment for Rockwood Type III Acromioclavicular Joint Dislocations? Clin Orthop Relat Res. 2023 May 1;481(5):1008-1013. doi: 10.1097/CORR.0000000000002545. Epub 2023 Jan 13. No abstract available. PMID 36728233